CLINICAL TRIAL: NCT01448239
Title: Injection Site Tolerability, Safety, Pharmacokinetics and Pharmacodynamics Study After a Single Dose Subcutaneous Treatment of Alirocumab SAR236553 (REGN727)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKD12010; U1111-1118-2935 (Other: UTN)
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2012-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- alirocumab SAR236553 (REGN727) - Dose A (Experimental): A single subcutaneous injection of Dose A
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) - Dose B (Experimental): A single subcutaneous injection of Dose B
  Interventions: Drug: alirocumab SAR236553 (REGN727)

INTERVENTIONS:
Drug: alirocumab SAR236553 (REGN727) — Pharmaceutical form:Solution Route of administration: Subcutaneous
  Arms: alirocumab SAR236553 (REGN727) - Dose A
Drug: alirocumab SAR236553 (REGN727) — Pharmaceutical form:Solution Route of administration: Subcutaneous
  Arms: alirocumab SAR236553 (REGN727) - Dose B

SUMMARY:
Primary Objective:

Injection Site Tolerability

Secondary Objectives:

* To assess the safety profile of alirocumab SAR236553 (REGN727)
* To assess the pharmacokinetic-pharmacodynamic relationship of alirocumab SAR236553 (REGN727)

DETAILED DESCRIPTION:
The total duration of study for each subject is up to 15 weeks including a screening period up to 3 weeks.

ELIGIBILITY:
Inclusion criteria:

* Serum troponin I level should not exceed the upper laboratory limit of normal.
* Male or female subject, between 18 and 65 years inclusive.
* Body weight between 50.0 and 95.0 kg inclusive if male, between 40.0 kg and 85.0 kg inclusive if female, body mass index (BMI) between 18.0 and 30.0 kg/m² inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 10 minutes resting in supine position.
* Normal standard 12-lead ECG after 10 minutes resting in supine position.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects
* If female, subject must use a double contraception method, except if she is sterilized for more than 3 months or postmenopausal.
* Serum LDL-C levels>100 mg/dL at screening visit.

Exclusion criteria:

* Subjects indicated for the use of statins according to criteria in National Cholesterol Education Program adult treatment panel III Guidelines, as updated in 2004 (see Appendix C).
* Initiation of a new diet or major change to a previous diet within 4 weeks prior to Screening (Day -21 to -2). Subjects must be willing to maintain a consistent diet for the duration of the study.
* Use of a medication or nutraceutical in order to alter serum lipids within 4 weeks prior to screening (Day -21 to -2), including but not limited to statins, ezetimibe, fibrates, niacin, or omega-3 fatty acids, bile acid resins.
* Fasting serum triglycerides >200 mg/dL measured after an 8 to 12 hour fast.
* History of a hypersensitivity reaction to doxycycline or similar compound.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pain using present pain intensity (PPI) verbal questionnaire | 6 weeks
Erythema at injection site by measuring diameter and qualitative assessment | 6 weeks
Edema at injection site by measuring diameter and qualitative assessment | 6 weeks

SECONDARY OUTCOMES:
Assessment of PK parameter - time to maximum concentration (tmax) | Up to 12 weeks
Assessment of PK parameter - maximum concentration (Cmax) | Up to 12 weeks
Assessment of PK parameter - area under curve (AUC) | Up to 12 weeks
Assessment of PK parameter - cluster of differentiation (CD) biomarker (CD29) | Up to 12 weeks
Assessment of PK parameter - terminal elimination half-life (t1/2z) | Up to 12 weeks
Pharmacodynamics: Change in LDL-C from baseline | Up to 12 weeks
Number of participants with Adverse Events | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States